CLINICAL TRIAL: NCT02476786
Title: Endocrine Treatment Alone as Primary Treatment for Elderly Patients With Estrogen Receptor Positive Operable Breast Cancer and Low Recurrence Score
Brief Title: Endocrine Treatment Alone for Elderly Patients With Estrogen Receptor Positive Operable Breast Cancer and Low Recurrence Score
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201611010
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cancer of Breast; Breast Neoplasms; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Anastrozole; exemestane; Fulvestrant; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endocrine therapy alone (Experimental): * Neoadjuvant endocrine therapy will be given at the discretion of the treating physician as directed by the package insert and could include the following: goserelin, anastrozole, letrozole, exemestane, fulvestrant, or tamoxifen
  * Frequency of office visits will be decided by the treating physician but must occur no less frequently than every 3 to 6 months for tumor assessment
  * After 6 months and after 12 months, patients will be assessed; patients who progress will have standard care recommended , and at any point a patient can opt to receive standard care even if she has not progressed on neoadjuvant endocrine therapy
  * Information on quality of life will be collected at baseline, Year 1, and Year 2 by the FACT-B questionnaire
  * Archival tissue will be collected and sent to Genomic Health for analysis using the Oncotype DX assay. The Recurrence Score predicts chemotherapy benefit and indicates the 10-year risk of recurrence (will not be used to determine treatment)
  Interventions: Behavioral: FACT-B; Drug: Goserelin; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Tamoxifen; Other: Archived tissue collection

INTERVENTIONS:
Behavioral: FACT-B — The FACT-B (Version 4) is a 37-item measure that contains the four general subscales along with the Breast Cancer-Specific subscale that assesses symptoms/concerns of particular relevance to breast cancer (e.g., body image, arm swelling and tenderness).
Drug: Goserelin
  Other Names: Goserelin acetate; Zoladex
Drug: Anastrozole
  Other Names: Arimidex®
Drug: Exemestane
  Other Names: Aromasin®
Drug: Fulvestrant
  Other Names: Faslodex®
Drug: Tamoxifen
  Other Names: Nolvadex®
Other: Archived tissue collection

SUMMARY:
Multiple neoadjuvant endocrine trials demonstrate that women with good prognosis tumors can be identified. These trials have also demonstrated that there are not adverse effects on overall outcome if women are treated with neoadjuvant endocrine therapy for several months prior to definitive treatment. A new standard of care needs to be defined for elderly women with good prognosis estrogen receptor (ER)+ tumors, since these women may benefit from endocrine therapy alone to treat their cancer without compromising local and distant control. The investigators hypothesize that endocrine therapy alone provides adequate local and systemic control of breast cancer in a subpopulation of women 70 or older with ER+ breast cancer and low Ki67 scores.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically or cytologically confirmed operable invasive breast cancer defined as cT1 or T2, N0-1, and M0.
* Disease must be ER+ and HER2-.
* Ki67 score/proliferative index ≤ 30% or low to intermediate mitotic index
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) by ultrasound or mammogram.
* 70 years of age or older.
* ECOG performance status ≤ 3
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior surgery for this cancer
* A history of other malignancy ≤ 5 years previous which would preclude endocrine treatment of their cancer.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the agents used in the study.
* Uncontrolled intercurrent illness as determined by their treating physician which would limit compliance with study requirements.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with endocrine therapies. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months
  * Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009].
  * In each RECIST response category Oncotype DX scores will be summarized with mean, standard deviation, minimum, 1st, 2nd (median) and 3rd quartiles, and maximum values. OncotypeDx scores range from 0 to 100, with scores <18 indicating low risk.

SECONDARY OUTCOMES:
Breast cancer-specific survival | 6 months
Breast cancer-specific survival | 1 year
Breast cancer-specific survival | 2 years
Rate of overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Aft, M.D, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu